CLINICAL TRIAL: NCT03847480
Title: Dose Painting of Head and Neck Cancer - The RADPAINT Pilot Study
Brief Title: Dose Painting of Head and Neck Cancer
Acronym: RADPAINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Einar Dale, Senior Consultant, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/398
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: Dose painting; 18F-FDG; Positron emission tomography; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose painting (Experimental): Dose painting
  Interventions: Radiation: FDG-PET guided dose painting

INTERVENTIONS:
Radiation: FDG-PET guided dose painting — The radiation dose inside the gross tumor volume is increased according to the voxel intensity (SUV - standardized uptake value) of pre-treatment FDG PET.

SUMMARY:
Dose-painting may increase the chance of cure at minimised radiation-induced toxicity in volumetric-arc radiotherapy (VMAT) for head and neck cancer. This trial (RADPAINT) investigates the safety of FDG-PET guided radiotherapy using VMAT dose-painting by contours for patients with head and neck cancer of poor prognosis.

DETAILED DESCRIPTION:
In this study, radiotherapy is planned using 18F-FDG PET/CT (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography) making one experimental "dose-painting by contours" SIB (simultaneous integrated boost) plan with a maximum point dose of 83 Gy. The participants will be given 73 Gy and 78 Gy minimum doses to two GTVs (gross tumor volumes inside the conventional GTV (68 Gy). GTV_73Gy and GTV_78Gy are determined from the SUV (standardized uptake values) from the 18F-FDG PET/CT according to the formula proposed by the Ghent group (Van der Straeten et al, R&O -06). It is expected to keep the level of normal tissue side-effects within or slightly above the level of conventional radiotherapy (i.e. maximum dose of 68 Gy).

In addition to the routine follow-up, the participants will be examined with 18F-FDG PET/CT (3 months after treatment and toxicity scoring at 6 weeks, 6 months, 1 year, 1.5 years and 3 years after radiotherapy (in addition to the routine follow-up).

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically verified invasive squamous cell carcinoma of the head and neck region; Oral cavity, hypopharynx cancer, larynx cancer and HPV ((human papillomavirus) negative oropharyngeal cancer.

Patients planned for standard curative treatment (radical radiotherapy with or without concomitant chemotherapy, with nimorazole hypoxic cell radiosensitizer)

Planned treatment at the Oslo University Hospital

Age > 18 years

WHO (World Health Organization) performance status 0-2

Exclusion Criteria:

TNM (primary tumor, regional nodes, metastasis) stage cT1 cN0-N1 cM0

Glottic cancer cT1-T2 cN0 cM0

HPV positive oropharyngeal carcinoma

Cancer in the soft palate

Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Late toxicity - mucosal ulcer | 1 year
  The study will be stopped if ≥ 2 patients experience mucosal ulcers grade ≥ 3 (CTCAE v 3.0/v4.0) without healing within the first year after radiotherapy. This endpoint will be assessed by clinical examination.
Acute or late toxicity | 1 year
  Any life-threatening toxicity (CTCAE v4.0) related to radiotherapy. This endpoint will be assessed by clinical examination.

SECONDARY OUTCOMES:
Acute toxicity | < 3 months after radiotherapy
  CTCAE v4.0
Late toxicity | 1 year
  CTCAE v4.0
Loco-regional control | 3 years
  FDG PET/CT at 3 months. Imaging thereafter if clinical progression.
Disease free survival | 3 years
  FDG PET/CT at 3 months. Imaging thereafter if clinical progression.
Overall survival | 3 years
  Date from central registry.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD PhD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Evensen ME, Furre T, Malinen E, Londalen AM, Dale E. Mucosa-sparing dose painting of head and neck cancer. Acta Oncol. 2022 Feb;61(2):141-145. doi: 10.1080/0284186X.2021.2022200. Epub 2022 Jan 6. No abstract available. PMID 34991431